CLINICAL TRIAL: NCT05235308
Title: Predictive Factors on the Results of Percutaneous Epidural Adhesiolysis in Patient With Chronic Spinal Pain
Brief Title: Predictive Factors on the Results of Epidural Adhesiolysis in Patient With Chronic Spinal Pain
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal investigator, Diskapi Teaching and Research Hospital
Other Study IDs: 127/22
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous adhesiolysis — Percutaneous adhesiolysis is a minimally invasive technique which involves the use of a spring-wound catheter, ideally placed in the ventrolateral aspect of the epidural space for the lysis of adhesions.

SUMMARY:
The primary aim of this exploratory study was to determine the demographic, clinical, and technical factors associated with treatment outcome, to create a better select treatment candidates.

ELIGIBILITY:
Inclusion Criteria:

* patients in whom percutaneous epidural lysis of adhesions was performed

Exclusion Criteria:

* nonadhesiolytic procedure
* lack of follow-up
* incomplete outcome data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with low back or leg pain who have not had positive responsive to the conservative treatments or procedures, such as epidural steroid injections.
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
pain intensity | baseline to 12 months post-procedure
  The visual analog scale is a numerical scale from 0 to 10; with 0 representing no pain and 10 representing the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No